CLINICAL TRIAL: NCT06044753
Title: Comparing the Effectiveness of Virtual Reality Versus Control Group in Reducing Preoperative Anxiety in Pediatric Patients
Brief Title: Comparing the Effectiveness of Virtual Reality in Paediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Maryam Budiman, Doctor, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JEP-2020-363
Record Dates: First submitted 2021-07-18; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Population; Preoperative Anxiety
Keywords: Induction of anaesthesia; Preoperative anxiety; Virtual reality; Paediatric patients

STUDY DESIGN:
Intervention Model Description: Paediatric Patients age 4 to 12 .
Who Masked: Participant
Masking Description: Masking of parents and patients, until entering the operation theatre
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm( Arm1) (No Intervention): Arm1 which is standard care/control group (as per usual practice). May use the distraction, Parental presence, or with musics, soft prep talks, distractions with toys, as per anaesthetist's usual practice.
  Patients will receive 100% oxygen of 6 L/min flow for 30 seconds. Nitrous oxide of 2 L/min will be added with ratio oxygen and nitrous oxide of 3:1. Sevoflurane inhalation will be initiated with 4% concentration for 30 seconds, followed by 8%. The induction will be proceeded in usual manner
- VR ( Virtual Reality) ( Arm2) (Experimental): Group 2 patients will choose one of the three YouTube videos, either Frozen theme song, SpongeBob or Minions according to their preference. The selected video will be played on the doctor's handphone and slotted into the VR headset.A handphone playing YouTube videos (either Frozen or SpongeBob or Minions VR cartoons) will be slotted into the VR headset prior to applying on the patient. They will have mask on first followed by the VR headset.
  Patients will receive 100% oxygen of 6 L/min flow for 30 seconds. Nitrous oxide of 2 L/min will be added with ratio oxygen and nitrous oxide of 3:1. Sevoflurane inhalation will be initiated with 4% concentration for 30 seconds, followed by 8%. The induction will be proceeded in usual manner
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Non immersive VR experience basically means providing a near reality environment for viewers, however, viewers won't be able to make any changes to it as they can only watch.
  This Non-immersive Virtual reality experience will be applied unto the child by using a headset that incorporates a computerized dimensional environment which will be simulated to make the child feel near reality .The VR headset consist of a cover for handphone slot, screen display, two lenses with adjustable eye pieces to focus, foam padding and adjustable elastic head mount strap.
  Arms: VR ( Virtual Reality) ( Arm2)

SUMMARY:
To the best of our knowledge,the investigators found only a study using VR in reducing preoperative anxiety in paediatric population. Ryu et al found that children who received preoperative VR tour of the operation theatre had perfect score in induction compliance checklist (ICC).

With these encouraging data,the investigators decide to conduct a study to determine whether the use of cartoon video VR headset during induction of anaesthesia is able to reduce preoperative anxiety and increase compliance during inhalation induction in children undergoing surgery.

DETAILED DESCRIPTION:
Patients will be reviewed prior to surgery, where explanation will be given and consent from patient's parents will be obtained. Once the parents consented for the study, patient will be recruited. Randomization will be carried out using a computer-generated system randomizing patient to two groups, Group 1 which is standard care/control group (as per usual practice) whereas Group 2 is VR intervention group. No premedication prescribed to patients.

Non immersive VR experience basically means providing a near reality environment for viewers, however, viewers won't be able to make any changes to it as they can only watch.

This Non-immersive Virtual reality experience will be applied unto the child by using a headset that incorporates a computerized dimensional environment which will be simulated to make the child feel near reality .The VR headset consist of a cover for handphone slot, screen display, two lenses with adjustable eye pieces to focus, foam padding and adjustable elastic head mount.

Group 2 patients will be tested for the suitability of mask size and applied together with the VR headset, meanwhile the strap for VR headset is adjusted accordingly to patient's head circumference and fixed for later use. The patient will choose one of the three YouTube videos, either Frozen theme song, SpongeBob or Minions according to their preference. These VR cartoon videos are 3-Dimension cartoon which are available to view for free. Frozen is a famous Disney cartoon, SpongeBob is an American animated cartoon series whereas Minions is an animated comedy film. The selected video will be played on the doctor's handphone and slotted into the VR headset. The codes for the VR cartoon videos will be scanned by the anaesthesiology trainees' registrars and specialists and downloaded into their handphone. The VR cartoon will be shown to the patients for 30 seconds to accustom them to wear the VR.

On the operation day, patients will enter the operation room as routine, while the primary investigator observes the patient and score their anxiety level using modified Yale Preoperative Anxiety Scale (mYPAS) upon arrival to operation room. Modified Yale Preoperative anxiety scale has been proved to be a reliable assessment tool. The mYPAS is a 22-itemized score divided into 5 categories which are activities, vocalization, expressing emotions, state of arousal and interaction with family members. Each category was scored from 1 to 4, except for vocalization, which scored from 1 to 6. As each category is itemized differently, partial weights were calculated and then added to the total score. The total score will be calculated post-intubation. The scoring will be done by dividing each item rating by the highest possible rating (i.e., 6 for the "vocalizations" item and 4 for all other items), the produced values will be summed. Divide by 4 and multiply by 100. mYPAS scores of ≤30 is described as non-anxious, and mYPAS score > 30 is described as anxious with the minimum score of 23.3 to maximum score of 100.13 Subsequently, the patients will be placed either on the operation table or be sited on the parent's lap depending on the patient's cooperation. The position of patients during induction is documented. Oxygen saturation probe will be applied on them. Baseline heart rate (HR) and SpO2 will be documented. Group 1 patients will receive standard care of inhaling gaseous induction through mask. For Group 2, a handphone playing YouTube videos (either Frozen or SpongeBob or Minions VR cartoons) will be slotted into the VR headset prior to applying on the patient. They will have mask on first followed by the VR headset. Patients in both groups will receive 100% oxygen of 6 L/min flow for 30 seconds. Nitrous oxide of 2 L/min will be added with ratio oxygen and nitrous oxide of 3:1. Sevoflurane inhalation will be initiated with 4% concentration for 30 seconds, followed by 8%. The induction will be proceeded in usual manner. Non-invasive blood pressure (NIBP) cuff and electrocardiogram (ECG) leads will be applied to the patients. BP, HR, SpO2 during induction and post-intubation will be recorded.

Following intubation, the attending anaesthetist will score the induction compliance checklist (ICC) which is an observational scale on the patient compliance to inhalational induction and mask acceptance. The ICC is a validated checklist and contains 10 negative behavioural groupings. The ICC score represents the sum of the groupings checked as present during induction; high scores correlate with poor behavioural compliance. A perfect induction (no negative behaviours) is scored as 0; the highest possible score is 10. For purposes of analysis, ICC scores were stratified into three categories: perfect (ICC = 0), moderate (1-3) and poor (≥4).

Anaesthetist in Group 2 will fill up a System Usability Scale (SUS). This scale was created by John Brooke in 1986 and used extensively to test numerous products and services. The SUS consists of 10 questions with 5 responses for each question ranging from "strongly agree" to "strongly disagree". The calculation of the usability score for SUS is, for each of the odd numbered questions, subtract 1 from the score. For each of the even numbered questions, subtract their value from 5. The produced values will be summed and multiply by 2.5. Questions 1,3,5,7 and 9 are positive whereas questions 2,4,6,8 and 10 are negative. The score is graded to five grades, score >80.3 (Grade A/ excellent), 68-80.3 (Grade B/ good), 68 (Grade C/ okay), 51-68 (Grade D/ poor) and ˂51 (Grade F/ awful).

In a situation where patient is unable to wear VR headset, the patient will be considered dropped off from the study. However, if the patient removes the VR headset or pushes away the mask during inhalation, data will still be recruited and considered, hence not a drop out case.

Collected data will be used to measure the association of mYPAS anxiety score with the ICC, which will determine the compliancy of patient to mask acceptance during induction. If the VR group shows a high mYPAS score yet a perfect or low ICC score compared to standard care group, hence the investigators can prove that VR does effectively decrease anxiety in paediatrics during inhalational induction.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) I or II patients.
2. Patients between 4-12 years of age.
3. Elective and emergency cases

Exclusion Criteria:

1. Maxillofacial anomalies
2. Skull anomalies that make fitting mask difficult
3. Visual and hearing impairment
4. Epilepsy
5. Contraindication to nitrous oxide and sevoflurane inhalation induction. For example; malignant hyperthermia, ear surgery and pneumothorax.
6. Autism spectrum disorder

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Compare Effectiveness of Virtual reality intervention versus standard care in reducing anxiety in paediatric patients undergoing inhalation induction | 1 year
  Primary objective is to compare effectiveness of virtual reality ( VR) intervention versus standard care in reducing anxiety of paediatric patients undergoing inhalation induction of anaesthesia by using the induction compliance checklist and compare with their mYPAS score. If the mYPAS score is high in Virtual Reality arm, however, Induction Compliance checklist is perfect score, hence we can conclude that VR arm patient have benefitted from the use of VR in reducing preoperative anxiety.

SECONDARY OUTCOMES:
Secondary objective is to investigate system usability of using virtual reality in inducing paediatric patients. | 1 year
  By using the system usability scale scoring by operators in virtual reality arm, we can determine whether the use of virtual reality headset is helpful in our daily clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Budiman, Principal Investigator — Universiti Kebansaan Malaysia
Locations (1):
- Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Ryu JH, Park SJ, Park JW, Kim JW, Yoo HJ, Kim TW, Hong JS, Han SH. Randomized clinical trial of immersive virtual reality tour of the operating theatre in children before anaesthesia. Br J Surg. 2017 Nov;104(12):1628-1633. doi: 10.1002/bjs.10684. Epub 2017 Oct 4. PMID 28975600
- [Background] Mifflin KA, Hackmann T, Chorney JM. Streamed video clips to reduce anxiety in children during inhaled induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1162-7. doi: 10.1213/ANE.0b013e31824d5224. Epub 2012 Oct 9. PMID 23051880
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388
- [Background] Malloy KM, Milling LS. The effectiveness of virtual reality distraction for pain reduction: a systematic review. Clin Psychol Rev. 2010 Dec;30(8):1011-8. doi: 10.1016/j.cpr.2010.07.001. Epub 2010 Jul 13. PMID 20691523